CLINICAL TRIAL: NCT05129501
Title: The Impact of an Adapted Version of the Strengthening Families Program on Reducing IPV Among Caregivers and ACEs Among Their Children (RCS Update)
Brief Title: The Impact of an Adapted Version of the Strengthening Families Program on IPV Among Caregivers and ACEs Among Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska Lincoln (Other)
Collaborators: Bennington College (Unknown); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21287
Record Dates: First submitted 2021-10-07; First posted 2021-11-22 (Actual); Results first posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Adverse Childhood Experiences; Domestic Violence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment: Tiwahe Wicaghwicayapi (Experimental): Part 1: Conduct informed consent process, perform baseline assessments (time 1 survey) Part 2: Complete the program over 7 weeks, fidelity checking during program Part 3: Takes survey immediately after program (time 2 survey) Part 4: Time 3 survey six months after Time 2 survey.
  Note: Participants are "randomized at the family level" into one of two arms (treatment or control), and children are assigned to the same arm as their caregiver.
  Interventions: Behavioral: Experimental
- Wait List Control: Tiwahe Wicaghwicayapi (No Intervention): Part 1: Conduct informed consent process, perform baseline assessments (time 1 survey) Part 2: Waitlist with access to resources while treatment group completes program Part 3: Takes survey immediately after experimental group completes program (time 2 survey) Part 4: Time 3 survey six months after Time 2 survey
  *Complete program.
  Note: Participants are "randomized at the family level" into one of two arms (treatment or control), and children are assigned to the same arm as their caregiver.

INTERVENTIONS:
Behavioral: Experimental — The Tiwahe Wicagwicayapi seven-session program is for children ages 10 to 14 who are Native American and/or living in poverty and their caregivers. The program begins with a traditional Lakota meal followed by family time and break-out time for caregivers only and children only. The program includes skill-building activities as well as the integration of Lakota language, history, and culture. The program is facilitated by diverse individuals, predominantly Native Americans in Rapid City and surrounding tribal communities.
  Arms: Treatment: Tiwahe Wicaghwicayapi

SUMMARY:
Adverse childhood experiences (ACEs) are unfortunately common and the known outcomes are concerning. However, very little is currently known about programs that may prevent ACEs among children, such as witnessing intimate partner violence (IPV) experienced by their caregivers. The purpose of this project is to adapt an existing evidence-based program (i.e., Strengthening Families) to prevent ACEs. A randomized control will be used to determine the initial efficacy of the program. The Strengthening Families program has demonstrated effectiveness in reducing substance use and initiation among youth, and some preliminary evidence suggests that it may be effective at reducing child maltreatment as well. Further, the Strengthening Families program promotes family bonding and cohesion, which are protective factors against ACEs. The Strengthening Families program has been adapted by researchers at UNL (Devan Crawford and Les Whitbeck) for Native American Families (i.e., BII-ZIN-DA-DE-DAH [Listening to One Another]) to prevent substance abuse. Using the Strengthening Families and BII-ZIN-DA-DE-DAH programs, the investigators seek to adapt these programs to prevent ACEs among youth ages 10-14 and their caregivers. The program adaptations are being led by a Community Advisory Board as well as community practitioner partners. The community has named the program Tiwahe Wicaghwicayapi (Lakota for: to strengthen/improve families). Native children and/or children living in poverty, ages 10 to 14, will participate in the program with their families. Participants will be "randomized at the family level" into one of two arms (treatment or control), and children were assigned to the same arm as their caregiver. Half of the families will go first and then the second half of the families will get the program after the last survey. The investigators will use surveys to see if and how the program is working and also interview some people who go through the program. A community Advisory Board is involved in all stages of this project and have the ultimate say about how data are shared.

DETAILED DESCRIPTION:
Research documents the concerning rates and negative outcomes of adverse childhood experiences (ACEs). ACEs include child abuse as well as indicators of household (e.g., exposure to intimate partner violence [IPV]) and neighborhood (e.g., community violence) dysfunction. To date, little is known about two-generation programs that may simultaneously prevent ACEs among children, including IPV in their caregivers. The purpose of the proposed project is to test the impact of a widely researched alcohol and drug abuse prevention program, the Strengthening Families Program (SFP), on reducing IPV among caregivers, child abuse, and other ACEs among their children (ages 10 to 14). The SFP is for both caregivers and children and consists of parenting skills, children's life skills, and family skills courses taught together in seven 2-hour group sessions preceded by a meal that includes informal family practice time and group leader coaching. Guided by social learning and ecological theories that emphasize the importance of the proximal family environment, the members of this multistakeholder collaborative believe that the SFP has the strong potential to be effective in reducing IPV in caregivers and additional ACEs in their children (e.g., child abuse) given that the SFP focuses on reducing myriad risk and protective factors for not only drug use but also for ACEs, including IPV.

To bolster the program's effectiveness, the investigators will adapt the SFP (the adapted program will be called Tiwahe Wicaghwicayapi, Lakota for "to strengthen/improve families") to be culturally relevant given the large presence of American Indians in Rapid City, SD, where the project will take place; and to have utility for a broader, diverse audience. Notably, service providers in racially diverse communities frequently do not have the resources to implement various prevention programs. Thus, there is a need in many communities for ACEs prevention programming that is culturally grounded and generalizable to the broader community. The investigators will further enhance the Tiwahe Wicaghwicayapi program to include additional evidence-based IPV prevention strategies (e.g., economic empowerment) for adults and peer-to-peer violence prevention strategies (e.g., bystander intervention) for youth.

Outcome and Process Evaluation Aim: To gather efficacy data of the Tiwahe Wicaghwicayapi program using a randomized control trial in which eligible families will be randomly assigned to the treatment condition or a wait-list control condition, using pre-, immediate post- and 6-month post- follow-up surveys to test for reductions in ACEs (e.g., child abuse) in youth ages 10 to 14 and reductions in IPV in caregivers for individuals in the treatment group compared to the wait-list control group. Participants will be "randomized at the family level" into one of two arms (treatment or control), and children are assigned to the same arm as their caregiver. Additionally, some outcome measures are collected only for the children or only for the caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Youth must be aged 10 to 14
* Must identify as a Native American, American Indian, Indigenous, and/or Lakota/Nakota/Dakota youth AND/OR live in poverty
* For caregivers, the inclusion criteria is that they must be a primary caregiver (e.g., parent, grandparent, etc) of a youth that meets criteria
* Both the youth and the caregiver(s) must be present to participate

Exclusion Criteria:

* Youth younger than 10 or older than 14
* Not identifying as Native American, American Indian, indigenous, and/or Lakota/Nakota/Dakota youth OR living in poverty
* Not being a primary caregiver of a youth that meets criteria
* Not having both the caregiver and youth present

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2021-10-09 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katie M Edwards, PhD, Principal Investigator — University of Nebraska Lincoln
Locations (1):
- Rapid City Family Project Office, Rapid City, South Dakota, United States

IPD SHARING:
Plan to Share IPD: No
This data will not be shared publicly due to the sensitive nature and history of data being used to oppress Indigenous groups. The Data Safety Monitoring Board and IRB has have the right to see deidentified data. Any publicly disseminated findings will be approved by the Native Advisory Board and surrounding tribal communities.

REFERENCES:
- [Background] Kumpfer, K. L. (1998). Prevention Interventions: The Strengthening Families Program. Drug Abuse Prevention Through Family Interventions, 160-207.
- [Result] Kaufman, E. A., Xia, M., Fosco, G., Yaptangco, M., Skidmore, C. R., & Crowell, S. E. (2016). The Difficulties in Emotion Regulation Scale Short Form (DERS-SF): Validation and replication in adolescent and adult samples. Journal of Psychopathology and Behavioral Assessment, 38(3), 443-455.
- [Result] Olson, D. H., Portner, J., & Bell R. Q. (1982). FACES II: Family adaptability and cohesion evaluation scales. Family Social Science, University of Minnesota, St. Paul, Minnesota.
- [Result] Small, S. A., & Kerns, D. (1993). Unwanted sexual activity among peers during early and middle adolescence: Incidence and risk factors. Journal of Marriage and the Family, 941-952.
- [Result] Straus, M. A., Hamby, S. L., Boney-McCoy, S., & Sugarman, D. B. (1996). The revised conflict tactics scales (CTS2) development and preliminary psychometric data. Journal of family issues, 17(3), 283-316.
- [Derived] Waterman EA, Wheeler L, Edwards KM, Herrington R, Mullet N, Hopfauf S. Measures to Assess Efficacy of Family-Based Programs for Indigenous Populations: Adaptation, Psychometric Properties, and Congruence. Fam Process. 2026 Mar;65(1):e70118. doi: 10.1111/famp.70118. PMID 41641935

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Tiwahe Wicaghwicayapi: Part 1: Conduct informed consent process, perform baseline assessments (Time 1 survey) Part 2: Complete the program over 7 weeks, fidelity checking during program Part 3: Takes survey immediately after program (Time 2 survey) Part 4: Time 3 survey six months after Time 2 survey.
  Experimental: The Tiwahe Wicagwicayapi seven-session program is for children ages 10 to 14 who are Native American and/or living in poverty and their caregivers. Participants were "randomized at the family" level into one of two arms (treatment or control). Randomized at the family level means that the caregiver was randomized into an arm, and then the rest of the family (that is, their children aged 10-14) were automatically assigned into that same study arm. Thus, caregivers and their children were always in the same arm (because it was a family intervention, the design demanded that the entire family be in the same study arm). The program begins with a traditional Lakota meal followed by family time and break-out time for caregivers only and children only. The program includes skill-building activities as well as the integration of Lakota language, history, and culture. The program is facilitated by diverse individuals, predominantly Native Americans in Rapid City and surrounding tribal communities.
- Wait List Control: Tiwahe Wicaghwicayapi: Part 1: Conduct informed consent process, perform baseline assessments (time 1 survey) Part 2: Waitlist with access to resources while treatment group completes program Part 3: Takes survey immediately after experimental group completes program (time 2 survey) Part 4: Time 3 survey six months after Time 2 survey.
  *Complete program.
  Note: Participants were "randomized at the family level" into one of two arms (treatment or control). Randomized at the family level means that the caregiver was randomized into an arm, and then the rest of the family (that is, their children aged 10-14) were automatically assigned into that same study arm. Thus, caregivers and their children were always in the same arm (because it was a family intervention, the design demanded that the entire family be in the same study arm).
Period: Overall Study
Arm/Group | Treatment: Tiwahe Wicaghwicayapi | Wait List Control: Tiwahe Wicaghwicayapi
Started | 173 (Number of participants including caregivers and children.) | 145 (Number of participants including caregivers and children.)
Additional Information: Number of Children Enrolled | 107 | 87
Additional Information: Number of Caregivers Enrolled | 66 | 58
Completed | 119 (Number of participants including caregivers and children. Within the 119 treatment participants who completed, 49 were caregivers and 70 were children.) | 104 (Number of participants including caregivers and children. Within the 105 control participants who completed, 43 were caregivers and 62 were children.)
Not Completed | 54 | 41
Not completed — Lost to Follow-up | 54 | 41

BASELINE CHARACTERISTICS:
Population: Number of participants, including both caregivers and children (all measures in this chart include both children and caregivers).
Groups:
- Treatment: Tiwahe Wicaghwicayapi: Part 1: Conduct informed consent process, perform baseline assessments (time 1 survey) Part 2: Complete the program over 7 weeks, fidelity checking during program Part 3: Takes survey immediately after program (time 2 survey) Part 4: Time 3 survey six months after Time 2 survey
  Experimental: The Tiwahe Wicagwicayapi seven-session program is for children ages 10 to 14 who are Native American and/or living in poverty and their caregivers. The program begins with a traditional Lakota meal followed by family time and break-out time for caregivers only and children only. The program includes skill-building activities as well as the integration of Lakota language, history, and culture. The program is facilitated by diverse individuals, predominantly Native Americans in Rapid City and surrounding tribal communities.
- Wait List Control: Tiwahe Wicaghwicayapi: Part 1: Conduct informed consent process, perform baseline assessments (time 1 survey) Part 2: Waitlist with access to resources while treatment group completes program Part 3: Takes survey immediately after experimental group completes program (time 2 survey) Part 4: Time 3 survey six months after Time 2 survey
  *Complete program
- Total: Total of all reporting groups
Arm/Group | Treatment: Tiwahe Wicaghwicayapi | Wait List Control: Tiwahe Wicaghwicayapi | Total
Number analyzed (Participants) | 173 | 145 | 318
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.09 (14.76) | 23.01 (15.71) | 22.55 (15.16)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Man/Boy | 61 | 45 | 106
  Woman/Girl | 104 | 92 | 196
  Other (e.g., Two Spirit) | 7 | 7 | 14
  Missing | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 147 | 119 | 266
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 6 | 1 | 7
  White | 1 | 7 | 8
  More than one race | 13 | 17 | 30
  Unknown or Not Reported | 5 | 0 | 5
Region of Enrollment [Number; unit: participants]
  United States | 173 | 145 | 318

OUTCOME MEASURES:

1. Primary Outcome: Adverse Childhood Experiences-Child Reported
Description: Comprehensive ACEs Measure (Higher scores indicate higher adverse childhood experiences). Note: As explained in the Pre-Assignment Details, participants were "randomized at the family level" into one of two arms (treatment or control), and children were assigned to the same arm as their caregiver. Additionally, some measures were collected only for the children or only for the caregivers. This particular measure was collected for children only.
Time Frame: Past 6 months
Population: This outcome measure is child-reported only.
Measure: Mean (Standard Deviation); unit: Mean number of adverse experiences
Arm/Group | Treatment: Tiwahe Wicaghwicayapi | Wait List Control: Tiwahe Wicaghwicayapi
Number analyzed (Participants) | 107 | 87
Mean number of adverse experiences | 2.48 (2.94) | 3.80 (3.56)

2. Primary Outcome: Conflict Tactics Scale-Adult Reported
Description: Intimate Partner Violence (Higher scores indicate higher levels of intimate partner violence victimization). Note: As explained in the Pre-Assignment Details, participants were "randomized at the family level" into one of two arms (treatment or control), and children were assigned to the same arm as their caregiver. Additionally, some measures were collected only for the children or only for the caregivers. This particular measure was collected for adults (i.e., caregivers) only.
Time Frame: Past 6 months
Population: This outcome measure is adult-reported only.
Measure: Mean (Standard Deviation); unit: mean number of IPV experiences
Arm/Group | Treatment: Tiwahe Wicaghwicayapi | Wait List Control: Tiwahe Wicaghwicayapi
Number analyzed (Participants) | 66 | 58
mean number of IPV experiences | 3.20 (5.10) | 2.21 (3.92)

ADVERSE EVENTS:
Time Frame: through study completion; that is, from baseline to six month follow-up
Arm/Group | Treatment: Tiwahe Wicaghwicayapi | Wait List Control: Tiwahe Wicaghwicayapi
All-Cause Mortality (participants affected / at risk) | 0/174 | 0/144
Serious Adverse Events (participants affected / at risk) | 0/174 | 0/144
Other Adverse Events (participants affected / at risk) | 0/174 | 0/144

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-11-15): https://cdn.clinicaltrials.gov/large-docs/01/NCT05129501/Prot_001.pdf
  • Statistical Analysis Plan (2021-10-22): https://cdn.clinicaltrials.gov/large-docs/01/NCT05129501/SAP_002.pdf